CLINICAL TRIAL: NCT07190365
Title: Goal-oriented Rehabilitation of Executive Functioning Using Video-telehealth to Improve Community Reintegration for Veterans With Chronic TBI and Cognitive Difficulties
Brief Title: Goal-oriented Telehealth Rehabilitation of Executive Functioning for Veterans With Chronic TBI
Acronym: GOALS TH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RRD1-001-24W; 1I01RD000680-01A2 (Other Grant/Funding Number: VA RRD)
Record Dates: First submitted 2025-09-05; First posted 2025-09-24 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Mild to Moderate Traumatic Brain Injury; Cognitive Rehabilitation; Veteran
Keywords: Mild to Moderate Traumatic Brain Injury; Cognitive Rehabilitation; Telehealth; Community Reintegration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinded assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GOALS TH (Experimental): The Goal-Oriented Attentional Self-regulation training involves ten 2-hour sessions of group-based telehealth training, three individual 1-hour telehealth training sessions, and approximately 20 hours of home practice. It is conducted in a small group format.
  Interventions: Behavioral: GOALS TH
- EDU TH (Active Comparator): The EDU TH training is an active control training matched with GOALS TH for therapist time, homework load, and participation in a group. It involves ten 2-hour telehealth sessions of group-based training, three individual 1-hour telehealth training sessions, and approximately 20 hours of home practice.
  Interventions: Behavioral: EDU TH

INTERVENTIONS:
Behavioral: GOALS TH — The Goal-Oriented Attentional Self-regulation training involves ten 2-hour sessions of group-based telehealth training, three individual 1-hour telehealth training sessions, and approximately 20 hours of home practice. It is conducted in a small group format.
  Arms: GOALS TH
Behavioral: EDU TH — The EDU TH training is an active control training matched with GOALS TH for therapist time, homework load, and participation in a group. It involves ten 2-hour telehealth sessions of group-based training, three individual 1-hour telehealth training sessions, and approximately 20 hours of home practice.
  Arms: EDU TH

SUMMARY:
Provision of interventions that address cognitive and emotional problems faced by Veterans with history of TBI pursuing community reintegration is an important concern for VA. Using telerehabilitation, the current project will help determine whether goal-directed training of attentional control functions via personally relevant activities will improve community integration for Veterans with history of TBI and cognitive difficulties. Findings may guide rehabilitation training towards providing services to maximize success in attaining complex functional goals in which Veterans can engage in skill strengthening 'where they are' (any location).

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) and comorbid conditions are prevalent in post-9/11 Veterans Chronic sequela of TBI can be highly debilitating due to deficits in the cognitive control processes, including attention, executive functions, and memory. Deficits in these cognitive control functions have been linked with difficulties in community reintegration, educational and occupational functioning, and are some of leading long-term disability causes among Veterans. As Veterans transition from military to community, many are interested in continuing to serve on the home front, with success in community, school, and work being essential to this goal.

At present, there are no validated evidence-based executive function tele-rehabilitation interventions to support community reintegration for Veterans with chronic TBI/Polytrauma. This study aims to increase access and availability of evidence-based, in-person administered cognitive rehabilitation training for Veterans with chronic TBI interested in improving their community integration. The adaptations include: 1) video telehealth delivery, and 2) focus on Veteran-chosen community integration goals,.

The objectives of this study are to investigate the feasibility and acceptability, as well as short (immediately post training), and longer-term (6 months post training) effectiveness of video telehealth cognitive rehabilitation training in 80 Veterans with history of chronic mild to moderate TBI and cognitive difficulties who are interested in improving their community integration. In a randomized, controlled intervention study, 80 Veterans with a history of mild to moderate TBI and residual cognitive difficulties will participate in telehealth GOALS and/or Brain Health Education - EDU interventions matched for time and intensity. Both groups will participate in pre and post training measurements at baseline and post training. Long-term follow-up will be at 6 months. Pre- and post-intervention and long term measurements will include performance on untrained: neuro-cognitive tests assessing targeted and non-targeted cognitive domains, individually defined goal attainment, and self-report measures of emotional regulation and daily functioning.

ELIGIBILITY:
Inclusion Criteria:

* History of mild to moderate TBI > 6 months ago
* Cognitive difficulties affecting daily functioning
* Age 18-65
* Veteran
* At least 12th grade education or equivalent * Interested in improving community reintegration

Exclusion Criteria:

* Amnesic/Severe memory problems
* Active Substance Abuse/Dependence
* Medical condition that may affect mental status/disrupt study participation
* Active psychotropic medication changes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2030-03-30 (Estimated); Study Completion 2030-03-30 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive performance -Overall Attention and Executive Function (AEF) Z score | Baseline, 10 week (post training), 6 month
  Performance on neurocognitive composite measure of attention and executive function post intervention vs control training will be assessed with Overall Attention and Executive Function (AEF) domain composite Z Score (calculated as the average of z scores of following tests: Letter Number Sequencing, Auditory Consonant Trigrams, Digit Vigilance, Trails B, DKEFS Stroop Inhibition, DKEFS Stroop Inhibition-Switching, DKEFS Verbal Fluency Switching, DKEFS Visual Fluency Switching). AEF Z score range is -3 to +3; higher score = better outcome.

SECONDARY OUTCOMES:
Functional outcomes - Mayo Portland Adaptability Inventory (MPAI) T score | Baseline, 10 week (post training), 6 month
  Performance on self-report measure of functional performance in daily life post intervention vs control training will be assessed with May Portland Adaptability Inventory (MPAI)- Total Score. MPAI Total T Score range is 20-80; higher score =worse outcome
Emotional regulation- Profile of Mood States (POMS) Z score | baseline, 10 week (post training), 6 month follow up
  Performance on self report measures of emotional regulation post intervention vs control training Overall psychological distress will be assessed with Profile of Mood States (POMS) questionnaire Total Mood Disturbance (TMD) Z Score. POMS Total Mood disturbance Z score range is -3 to +3; higher score = better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Tatjana Novakovic-Agopian, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No
Electronic datasets underlying publications will be de-identified and anonymized.
  Limited datasets without individually identifiable data will be maintained locally on VA protected servers until the appropriate data use agreements are in place.